CLINICAL TRIAL: NCT06172634
Title: A Single-center Clinical Study to Evaluate the Safety and Efficacy of Autologous Bone Marrow-derived DCs(CellgramDC-WT1) and Immune Checkpoint Inhibitors in Patients With Metastatic Pancreatic Cancer Who Have Failed First-line or More Standard Chemotherapy
Acronym: DICI_PC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jong-Ho Won, Soonchunhyang University Seoul Hospital, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC_ICI_PC_1
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pancreas Cancer
Keywords: dentritic cell; immune checkpoint inhibitors
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: dentritic cell + immunechekpoint inhibitor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC + ICI (Experimental)
  Interventions: Drug: dentritic cell infusion and immunecheckpoint inhibitor

INTERVENTIONS:
Drug: dentritic cell infusion and immunecheckpoint inhibitor — dentritic cell infusion and immunecheckpoint inhibitor

SUMMARY:
To evaluate the safety and effectiveness of immune cell therapy using autologous bone marrow-derived dendritic cells and immune checkpoint inhibitors in patients with metastatic pancreatic cancer who have failed at least one standard anticancer treatment.

DETAILED DESCRIPTION:
After a test subject agrees in writing to participate in a clinical study, if he or she is determined to fit the selection criteria and does not meet the exclusion criteria through a screening process, he or she is enrolled in the clinical study.

After consenting to the study, subjects set a bone marrow collection date within 7 days of registration, and granulocyte colony-stimulating factor (G-CSF) is administered the day before bone marrow collection. After bone marrow collection (approximately 30-50 ml) on the day of bone marrow collection, autologous bone marrow-derived dendritic cells (Cellgram-DC-WT1) made by isolating CD141+ cells from the bone marrow are administered intravenously together with pembrolizumab, at 3-week intervals. After repeating the test drug administration 3 times at 3-week intervals, a radiological response evaluation of the tumor is performed, and a decision is made to continue or terminate the test drug administration according to the response evaluation results. If the response evaluation results for the tumor fall into a complete response, partial response, or stable disease, administration of the test drug is continued, and the response evaluation is repeated three times at three-week intervals. If the response evaluation result for the tumor is progressive disease, administration of the test drug is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically confirmed to have pancreatic cancer and diagnosed as recurrent or metastatic
* Patients whose disease was confirmed to have progressed according to RECIST v1.1 after 1st or more standard anticancer treatments
* Patients satisfying systemic performance status ECOG 0-2
* Patients who have not undergone surgery, radiation therapy, or immunotherapy within 4 weeks and have recovered from side effects (However, tissue collection procedures that do not affect the test subject's condition are permitted at the discretion of the researcher.)
* Patients who voluntarily agreed in writing to participate in this clinical study

Exclusion Criteria:

* Patients with malignant tumors other than non-melanoma skin cancer in the past 3 years
* Patients who have previously received anti-tumor immunotherapy (anti-PD1, anti-PDL-1, or CTLA4 inhibitor, etc.) or participated in clinical studies related to immunotherapy or cell therapy
* Patients with active autoimmune disease requiring systemic immunosuppressive treatment
* Patients with a history of organ or hematopoietic stem cell transplantation
* Patients with acute or chronic infection requiring systemic treatment
* Other cases where the test manager determines that it is not suitable for clinical research

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
treatment related adeverse event | for 1yr

SECONDARY OUTCOMES:
overall response rate | for 1yr
  treatment response